CLINICAL TRIAL: NCT00907634
Title: Prospective Evaluation of Intrafractional and Interfractional Cervical Motion During External Beam Radiation for Intact Cervical Cancer by the Calypso® 4D Localization System™
Status: Withdrawn | Type: Observational
Why Stopped: Study closed by IRB because a Continuing Review and/or Close-Out have not been submitted.
  Study closed by IRB
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Peter J. Rossi, MD, Principal Investigator, Emory University
Other Study IDs: IRB00013078; EmoryCervicalMotion (Other: Other)
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Cervical Cancer
Keywords: cervix; cervical; radiation
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find out how the cervix normally moves during radiation treatment. This study will also evaluate how cervical cancer shrinks during chemotherapy and radiation. By better understanding these two things, the investigators can see if radiation could safely be given in a more focused way in the future.

The investigational portion of this study includes (1) daily cone beam CT scans to confirm transponder placement and evaluate tumor changes during treatment and (2) tracking movement of the cervix during daily radiation treatment.

DETAILED DESCRIPTION:
There has been recent interest in the use of Intensity Modulated Radiation Therapy (IMRT), a form of focal external beam radiation for intact cervical cancer. IMRT has been proposed as (1) an alternative treatment of the whole pelvis in an attempt to reduce the dose of radiation delivered to normal tissues and (2) a replacement for brachytherapy as an integrated or sequential radiation boost instead of intracavitary brachytherapy. At other tumor sites, IMRT has allowed for radiation dose escalation to the tumor while sparing adjacent normal tissues. IMRT requires greater accuracy of targeting and understanding of tumor and organ motion and tumor regression during radiotherapy to protect adjacent normal tissues and prevent against tumor underdosage.

Currently, there is limited knowledge of cervical organ motion. Previous studies have evaluated interfractional cervical motion [daily set-up variation, i.e. the location of the cervix on Day 1 vs. Day 2 or Day 30 of radiation treatment] with weekly CT and MRI scans or localization of fiducial markers evaluated by fluoroscopy daily before radiation therapy. There is no published literature regarding intrafractional cervical motion [motion during a single radiation treatment]. We propose a prospective clinical trial utilizing the Calypso® 4D Localization System™ to evaluate intrafractional and interfractional cervical motion for intact cervical cancer.

The Calypso® 4D Localization System™ is an FDA approved tumor localization system for adjunctive use in patients undergoing radiation therapy for prostate cancer. The system is designed to provide accurate, objective, and continuous 3-dimensional localization of the treatment target for patient alignment and target position monitoring relative to the isocenter of the linear accelerator. The Calypso system consists of implantable electromagnetic transponders, each with a unique resonant frequency. An array is placed over the patient and remains in place during radiation delivery. Source coils in the array emit electromagnetic signals that excite the transponders identifying the position of each individual transponder. The transponder position can be continuously monitored throughout treatment delivery reporting transponder motion in lateral, superior-inferior (SI), and anterior-posterior (AP) directions.

Our goal is to enroll 10 patients over a 1-2 year time period with intact cervical cancer (Stage IB-IVA) who will receive definitive radiation therapy at Emory University Hospital and Emory Crawford Long Hospital. Two Calypso beacons will be attached within a cervical "Smit" sleeve [1 superior, 1 inferior] which will be placed within the cervical os prior to CT simulation (radiation planning session). The cervical sleeve will be sutured in with 2 stitches. The location of the transponders will be tracked throughout the treatment delivery. Daily cone beam CT on the radiation treatment machine will also be utilized to confirm transponder placement and evaluate tumor volume changes during the treatment course. There will be no treatment field modifications based on cervical (transponder) displacement. While enrolled on this study, patients will be treated with the current standard of care treatment: 5 weeks of external beam radiation with concurrent weekly cisplatin and followed a focal radiation "boost" using intracavitary brachytherapy. The 5 weeks of external beam radiation therapy will be delivered with a conventional 4-field technique to the whole pelvis for a total of 45Gy at 1.8 Gy per fraction. All external beam radiation treatments will be delivered at the Emory Clinic, Clifton Road. The cervical sleeve will be removed following the external beam portion of therapy.

The calypso beacons will be provided free of charge for this study and there will be no additional costs to the patient or the Radiation Oncology Department for patients enrolling in this study. No additional risks are anticipated for patients enrolled in this study compared to the current standard of care treatment. The only "tests" that are part of our protocol that are outside of the standard of care for the treatment of intact cervical cancer would be the use of the (1) Calypso array used to localize the calypso "beacons" and (2) daily cone-beam CT scans to evaluate cervical cancer response to therapy. The Radiation Oncology department regularly uses both systems for patient set-up for other solid tumors and there will be no additional charge for these tests.

We believe this study will greater improve our current knowledge of cervical cancer motion and tumor regression during radiation therapy. There is concern that smaller radiation fields, as would be delivered with IMRT could underdose portions of the tumor resulting in inadequate local tumor control and compromising cure. As a result of this study will be able to infer if IMRT is a safe and reasonable treatment option for patients with intact cervical cancer. Knowledge of the extent and direction of cervical motion will also help determine IMRT treatment margins.

ELIGIBILITY:
Inclusion Criteria:

* Stage IB-IVA Cervical Squamous cell carcinoma
* Karnofsky Performance Score 60-100

Exclusion Criteria:

* Other histologies
* Karnofsky Performance Score < 60

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stage IB-IV Cervical cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossi, MD, Principal Investigator — Emory University